CLINICAL TRIAL: NCT04384016
Title: A Cross-over, Open-label, Single-group Study to Evaluate the Safety and Immunogenicity of Live Attenuated Varicella Vaccine Skyvaricella Injection (Inj.) Developed by SK Bioscience (Company Limited) Co., Ltd of South Korea in Healthy Volunteer Vietnamese Children From 12 Months to 12 Years Old
Brief Title: Safety and Immunogenicity of Skyvaricella Injection in Healthy Volunteer Vietnamese Children From 12 Months to 12 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Collaborators: Vabiotech (Industry)
Responsible Party: Principal Investigator, Pham Ngoc Hung, Principal Investigator, Vietnam Military Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VX.2019.08
Record Dates: First submitted 2020-05-02; First posted 2020-05-12 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Chickenpox
Keywords: Chickenpox; varicella-zoster virus; varicella vaccine
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluating the Safety of Skyvaricella Inj. (Experimental): The main target:
  • Evaluating the safety of Live Attenuated Varicella Vaccine SKYVaricella injection in healthy Vietnamese children from 12 months to 12 years, with a single injection
  Interventions: Biological: Skyvaricella Injection
- Evaluating the Immunogenicity of Skyvaricella Inj. (Experimental): Secondary target
  • Evaluating the immunogenicity of Live Attenuated Varicella Vaccine SKYVaricella injection in a small group of healthy Vietnamese children from 12 months to 12 years, with a single injection.
  Interventions: Biological: Skyvaricella Injection

INTERVENTIONS:
Biological: Skyvaricella Injection — The main target is evaluating the safety of SKYVaricella injection in healthy Vietnamese children from 12 months to 12 years, with a single injection.
  The secondary target is to Assess the immunogenicity of SKYVaricella inj. in a small group of healthy Vietnamese children from 12 months to 12 years, with a single injection.

SUMMARY:
This is a cross-over, open-label, single-group study. The study subjects were children 12 months to 12 years of age who will be vaccinated with a single dose. The duration of follow-up for safety evaluation and immunogenicity (on a small group) is 6 weeks (+ 2 weeks).

The main target:

• Evaluating the safety of live attenuated Varicella vaccine [Oka / SK], lyophilized powder and solvent for subcutaneous injection (SKYVaricella inj.) in healthy Vietnamese children from 12 months to 12 years, with a single injection.

Secondary target:

• Assess the immunogenicity of live attenuated Varicella vaccine [Oka / SK], lyophilized powder and solvent for subcutaneous injection (SKYVaricella inj.) in a small group of healthy Vietnamese children from 12 months to 12 years, with a single injection.

DETAILED DESCRIPTION:
The Safety of Skyvaricella Injection:

* The incidence of a chickenpox-like local rash (injection site) or chickenpox-like rash (disseminated) between 1 and 6 weeks after vaccination
* The incidence and severity of events (local and systemic) within 30 minutes after vaccination
* The incidence of expected systemic and local adverse events within 7 days after vaccination
* The incidence of serious adverse events and Unexpected adverse events within 6 weeks after vaccination The Immunogenicity of Skyvaricella Injection: seroconversion rate by Fluorescent antibody to membrane antigens (FAMA) test 6 weeks after investigational vaccination

ELIGIBILITY:
Inclusion Criteria:

* Children from full 12 months to full 12 years of age, healthy, agreed to participate by parents/guardians and allowed to monitor during the study period.
* The legal parent/guardian signs the study consent form, fully understanding the details of the study. Be fully explained and voluntarily agree to participate in the study and be able to follow the instructions provided by the study.
* The parent / legal guardian agrees in writing and is deemed to be able to cooperate with the study and meet all the requirements described in the protocol during the study.
* If girls are menstruating, a negative pregnancy test should be performed on the day of vaccination and consent to birth control practices within 3 months after vaccination.

Exclusion Criteria:

* Hypersensitivity reaction to any component of the research vaccine, such as gelatin or neomycin.
* Has been vaccinated against chickenpox before.
* History of chickenpox.
* People who have been exposed to chickenpox at home, day care, school, etc. within 4 weeks before getting the IP vaccine.
* Persons with acute or chronic cardiovascular disorders (CS) of clinical significance (respiratory, endocrine and neurological (including hematological diseases, leukemia), all types of lymphoma and other malignancies affecting the bone marrow or lymphatic system).
* People with a history of hypersensitivity to immunization, or Guillain-Barre syndrome.
* Patients who have used or are expected to use immunosuppressive or immunomodulatory therapies 6 months prior to the study vaccine up to 3 visits (6 + 2 weeks after vaccination) -xin) (e.g. chemotherapy drugs such as Cyclophosphamide, 6-Mercaptopurine, Azathioprine, Methotrexate, Cyclosporine A, Rapamycin and Leflunomide / biological treatments such as tumor necrosis factor [TNF-α], antiallergic drugs (antibodies, monoclonal antibodies and antisera / lymphocytes).
* Congenital or acquired immunodeficiency, lowering blood gammaglobulin and blood gammaglobulin disorder.
* Persons with a family history of congenital or hereditary immunodeficiency.
* Persons who live in the same household as a member of a high-risk group for varicella infection (for example, infants aged 0 to 4 weeks, pregnant women without a history of chickenpox vaccination and disease nuclear immunodeficiency factor).
* People currently suffering from tuberculosis.
* Ear canal temperature of 38.0 ° C or higher on the day of the vaccination.
* Those who received or expected to receive salicylate from 14 days before the IP vaccine to the 3rd visit (6 + 2 weeks after the IP vaccine).
* Persons who have received or are expected to receive human immunoglobulins, whole blood or blood-derived products such as packed red blood cells (RBC), intravenous immunoglobulins (IVIG) or globulins immunity to varicella zoster (VZIG) from 5 months prior to the IP vaccine to the 3rd visit (6 + 2 weeks after the IP vaccine).
* Persons who have received or are expected to receive other vaccines 4 weeks prior to the IP vaccine visit 3 (6 + 2 weeks after the IP vaccine).
* Those who received or expected to receive steroids from 3 months prior to the IP vaccine to the 3rd visit (6 + 2 weeks after the IP vaccine) (However, in the case of steroid use Low doses [eg <2 mg Prednison / kg / day up to a maximum of 20 mg / day for <2 weeks], the patient can participate in the study if use can be suspended until 3rd Visit after getting the IP vaccine).
* Persons who received or expected to receive antiretroviral drugs from 1 month prior to the IP vaccine to 3rd visits (6 weeks after vaccination + 2 weeks) during the clinical study period ( However, in the case of topical antiviral drugs, patients can participate in the study).
* People who received or expected to receive other IPs in another clinical study from 1 month before the IP vaccine to the 3rd visit (6 + 2 weeks after the IP vaccine).
* Others are considered ineligible to participate in research according to the researcher's judgment.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
the Safety of Skyvaricella Injection | between 1 and 6 weeks after vaccination
  The incidence of a chickenpox-like local rash (injection site) or chickenpox-like rash (disseminated).
the Safety of Skyvaricella Injection | within 30 minutes after vaccination
  The incidence and severity of events (local and systemic)
the Safety of Skyvaricella Inj. | within 7 days after vaccination
  The incidence of expected systemic and local adverse events
the Safety of Skyvaricella Injection | within 6 weeks after vaccination
  The incidence of serious adverse events and Unexpected adverse events

SECONDARY OUTCOMES:
the Immunogenicity of Skyvaricella Injection | 6 weeks after investigational vaccination
  seroconversion rate by Fluorescent antibody to membrane antigens (FAMA) test

CONTACTS AND LOCATIONS:
Overall Officials: Pham N Hung, As. Prof., Principal Investigator — Vietnam Military Medical University
Locations (1):
- CDC Ha Nam, Phủ Lý, Ha Nam, Vietnam

IPD SHARING:
Plan to Share IPD: No